CLINICAL TRIAL: NCT06339307
Title: A Prospective Clinical Study to Validate a Preoperative Risk Scoring Model for Lymph Node Metastasis in Gastric Cancer Patients
Brief Title: A Prospective Clinical Study to Validate a Preoperative Risk Scoring Model for LNM in GC Patients
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DJY004
Record Dates: First submitted 2024-03-17; First posted 2024-04-01 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2024-02

CONDITIONS: Predictive Cancer Model; Gastric Cancer; Lymph Node Metastasis
MeSH Terms: conditions — Stomach Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with LNM: Patients with gastric cancer who underwent curative gastrectomy and developed lymph node metastasis.
- without LNM: Patients with gastric cancer who underwent curative gastrectomy and did not develop lymph node metastasis.

SUMMARY:
In our prior research, a risk scoring model for the occurrence of lymph node metastasis in patients who underwent radical gastrectomy for gastric cancer was established. To further validate this scoring model, a prospective study has been designed with the aim of prospectively assessing the model's clinical applicability.

DETAILED DESCRIPTION:
The study was a single-centre, prospective study. Data prospectively accrued were employed to evaluate the concordance between observed patient outcomes, with respect to lymph node metastasis status post-curative gastrectomy, and the prognostications tendered by the established risk scoring model, thereby appraising the model's clinical applicability and validity.

ELIGIBILITY:
Inclusion Criteria:

1. Primary gastric adenocarcinoma;
2. Curative surgery (with R0 resection, excluding palliative surgery and cases with distant metastasis).

Exclusion Criteria:

1. Patients with autoimmune diseases, inflammation, or hematological disorders;
2. Patients with a history of or concurrent other cancers;
3. Presence of active infection and inflammation (based on WBC count, patients with count of 10×10^9 or higher should be evaluated through medical record examination for the presence of infection);
4. Active bleeding (as determined by endoscopic ultrasound and HGB ≤ 90);
5. Post neoadjuvant radiotherapy or chemotherapy;
6. History of blood transfusion, corticosteroid use, or leukocyte-stimulating medications within the past month prior to blood draw;
7. Incomplete clinical and pathological data.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with gastric cancer pathologically and underwent curative gastrectomy.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-04-21 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
lymph node metastasis | 1 month after curative surgery
  Collect postoperative pathological data from gastric cancer patients who have undergone curative gastrectomy to determine the occurrence of lymph node metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality, China

DOCUMENTS (3):
  • Study Protocol (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT06339307/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT06339307/SAP_001.pdf
  • Informed Consent Form (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT06339307/ICF_002.pdf